CLINICAL TRIAL: NCT06854926
Title: Effects of Helping Relationship from Significant Others in Patients with Hypertension Adhere to Healthy Lifestyles and Medication.
Brief Title: Helping Relationship from Significant Others in Patients with Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCKUH
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Hypertension; Significant Others
Keywords: hypertension; significant others; helping relationship; healthy lifestyles; medical adherence
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: patients with hypertension
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helper team (Experimental): Significant others of patient will practice strategies of helping relationship to help patients improve their health condition.
  Interventions: Behavioral: Helping relationship from significant others
- Usual team (Placebo Comparator): Patients of this team accept usual care
  Interventions: Behavioral: Usual team

INTERVENTIONS:
Behavioral: Helping relationship from significant others — Helping relationship from significant others is the intervention of this study. We will use four strategies, including warning mechanisms, target setting, encouragement, and feedback.
  Arms: Helper team
Behavioral: Usual team — Patients of this team accept usual care
  Arms: Usual team

SUMMARY:
The goal of this clinical trial is to learn if helping relationship from significant others in patients with hypertension improve the adherence to healthy lifestyles and medication. The main questions it aims to answer:

Does helping relationship from significant others improve in patients with hypertension the adherence to healthy lifestyles and medication? Is helping relationship from significant others helpful to patients with hypertension?

Researchers will compare helping relationship from significant others with routine care to see if the intervention works to improve hypertension.

Participants and their significant others will be participate in this study.

Significant others will prompt participants about:

Take the medicine according to the prescription. Sodium restriction Alcohol limitation Body weight reduction Cigarette smoke cessation Diet adaptation Exercise adoption

DETAILED DESCRIPTION:
With an increasing prevalence of Hypertension around the world, chronic disease management has become an optimal issue. There are many components about hypertension management, such as diet, exercise, medication adherence and social support. As the current pandemic situation and the shortage of healthcare providers, the patients must be aware of health condition themselves. We need more efficacious approaches to achieve better hypertension management. Due to the traditional methods can't lead to better disease management, social support might improve the blood pressure control and their poor adherence to treatment.

This study aims to develop helping relationship from significant others in Hypertension patients adhere to healthy lifestyles. We plan to recruit patients in southern Taiwan medical center. Those who aged 18 years and over, diagnosed hypertension, taking at least one western antihypertensive medication once a day and those who have significant others. The trial will conduct in a medical center as a quasi-experimental study. Patients will be divide into two groups. They will all recept the knowledge of Hypertension. The intervention group will receive another information about how they conduct their helping relationship as significant others. After intervention, we will compare the blood pressure, medication adherence, lifestyles and helping relationship between intervention and control groups. All data will be analyzed by using SPSS.

The helping relationship by significant others would be beneficial to hypertension management. Participants are willing to control their blood pressure and reveal more consideration for their health.

Chronic disease depends on not only self efficacy but also the whole family support. With helping relationship by significant others, we can adjust care plan according to individual needs. Hope to reach the goal of whole person care.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with Hypertension
* Patients with Hypertension those who accompanied with their significant other
* Clear consciousness and able to communicate with Mandarine or Taiwanese
* Willing to participate in this project
* Bring their own blood pressure monitor
* Currently taking at least one Western antihypertensive medication once/day

Exclusion Criteria:

* Without taking any medication of hypertension
* Acute medical issue
* Be diagnosed with Cognitive deficiency
* Currently join another research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 3 months
  Medication Adherence Scale is a reliable and valid measure of medication adherence in Taiwanese patients with hypertension. We will know the medication adherence of Taiwanese patients with hypertension by using the scale.
Health promotion lifestyle | 3 months
  Health promotion prevents illness, enhances wellbeing, and creates a healthy lifestyle at all stages of life.The HPLP developed by Walker and others in 1987 evaluates health promotion lifestyle related behaviours.
Helping Relationships From Significant Others | 3 months
  Using the helping relationships from significant others (HRSO) scale assists patients, in adopting a healthy lifestyle to decelerate disease progression, complications, and mortality.

SECONDARY OUTCOMES:
Blood pressure measurement | 3 months
  We will ask patients record blood pressure at home and compare with office blood pressure monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Syuan Huang, Study Chair — master's student
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided